CLINICAL TRIAL: NCT02769884
Title: Multiple Model Probabilistic Predictive Control (MMPPC) Outpatient Clinical Protocol
Brief Title: MMPPC Outpatient Clinical Protocol 2016
Acronym: MMPPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rensselaer Polytechnic Institute (Other)
Collaborators: Stanford University (Other); University of Colorado, Denver (Other); Mount Sinai Hospital, New York (Other)
Responsible Party: Principal Investigator, B. Wayne Bequette, Professor, Department of Chemical & Biological Engineering, Rensselaer Polytechnic Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMPPC- outpatient-2016
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Type 1 Diabetes
Keywords: artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Use the MMPPC system for 72 hours in a hotel setting
Oversight: Data Monitoring Committee: No

ARMS (1):
- MMPPC arm (Experimental): Subjects in this arm will wear the experimental MMPPC algorithm artificial pancreas for 72 hours in a hotel/house setting. The study period will involve unannounced meals and exercise
  Interventions: Device: MMPPC algorithm artificial pancreas

INTERVENTIONS:
Device: MMPPC algorithm artificial pancreas — An artificial pancreas system using the MMPPC algorithm, Roche insulin pump, and Dexcom CGM

SUMMARY:
This study trials a prototype artificial pancreas system that consists of a Roche insulin pump, a Dexcom continuous glucose monitor (CGM), and an experiential MMPPC (multiple model probabilistic predictive control) algorithm housed on an android cell phone. The system doses insulin based on CGM sensor glucose levels and the experimental algorithm.

The aim of this clinical study is to determine the efficacy of the MMPPC controller in adolescents and adults with type 1 diabetes in a hotel setting.

DETAILED DESCRIPTION:
This study trials a prototype artificial pancreas system that consists of a Roche insulin pump, a Dexcom continuous glucose monitor (CGM), and an experiential MMPPC (multiple model probabilistic predictive control) algorithm housed on an android cell phone. The system doses insulin based on CGM sensor glucose levels and the experimental algorithm. The algorithm runs through a glucose control platform called the DiAs (Diabetes Assistant)

The aim of this study is to determine the safety and feasibility of the MMPPC controller in adults and adolescents with type 1 diabetes testing the use of predefined tuning parameters to provide adaptability to patient. We will assess the safety of the system with both unannounced meals, and meals using a meal announcement with a premeal insulin bolus based on the subject's estimated carbohydrate content of the meal

ELIGIBILITY:
3.1 Eligibility Criteria

1. Clinical diagnosis of type 1 diabetes for at least 12 months 2. Daily insulin therapy for at least 12 months 3. Age between 15.0 to 55.0 years of age 4. Use of an insulin pump for at least 3 months 5. Current use of continuous glucose monitoring with Dexcom sensor 6. Subject comprehends English 7. Females of childbearing potential must use an adequate method of contraception and have a negative pregnancy test 8. Total daily insulin requirement ≥ 0.3 units/kg/day 9. A1C between 7.0 and 10% 3.2 Exclusion Criteria

1. Diabetic ketoacidosis in the past 6 months
2. Hypoglycemic seizure or loss of consciousness in the past 6 months
3. Hypoglycemia unawareness as defined by no recognition of hypoglycemia until the glucose is <60 mg/dL and no adrenergic symptoms at glucose of 60 mg/dL (shakiness, palpitations, diaphoresis). Subjects will also be administered the Clark questionnaire for hypoglycemia unawareness. If they have a score ≥ 4, they are excluded from the study
4. Subjects requiring an intermediate or long-acting insulin (such as NPH, detemir or glargine)
5. Subjects using other anti-diabetic medications other than insulin (oral or injectable) at the time of enrollment. Any prior use of other anti-diabetic medications must be washed out for at least 8 weeks prior to enrollment.
6. Current use of other medications, which in the judgment of the investigator would be a contraindication to participation in the study
7. Subject has a medical disorder that in the judgment of the investigator will affect completion of any aspect of the protocol
8. Subject is currently participating in another investigational device or drug study within 30 days or 5-half lives of the drug.
9. Subject has a history of any cardiac or vascular disorder including, but not limited to, myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, arrhythmia or thromboembolic disease
10. An EKG will be obtained on subjects who are ≥ 45 years of age, or who have had a 20 year history of diabetes and are ≥ 30 years of age. Subjects will be excluded if they have an abnormal EKG consistent with coronary artery disease or increased risk of malignant arrhythmia including, but not limited to, evidence of active ischemia, prior myocardial infarction, proximal LAD critical stenosis (Wellen's sign), prolonged QT interval (> 440 ms). Non-specific ST segment and T wave changes are not grounds for exclusion in the absence of symptoms or history of heart disease.
11. Subject has a history of hepatic disease
12. Subject has renal failure on dialysis
13. Systolic blood pressure > 160 mmHg on screening visit
14. Diastolic blood pressure > 90 mmHg on screening visit
15. Subjects with inadequately treated thyroid disease or celiac disease
16. Subject has a neurologic disorder that in the judgment of the investigator will affect completion of the protocol
17. Subject has received inpatient psychiatric treatment in the past 6 months
18. Subject consumes more than an average of 4 standard alcoholic drinks/day in the last 30 days
19. Subject has an active skin condition that would affect sensor placement
20. Subject is unable to avoid acetaminophen for the duration of the study
21. Subject consuming less than 100g of carbohydrates daily

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mean CGM glucose value | 72 hours
  Average CGm glucose value during the experimental trial
CGM percent time < 60 mg/dl | 72 hours
  Percent of time the CGM was reading <60 mg/dl

SECONDARY OUTCOMES:
CGM percent time < 50 mg/dl | 72 hours
  Percent of time the CGM was reading <50 mg/dl
CGM percent time < 70 mg/dl | 72 hours
  Percent of time the CGM was reading <70 mg/dl
% 70-140 mg/dl | 72 hours
  Percent of time CGM glucose levels were between 70-140 mg/dl
% 70-180 mg/dl | 72 hours
  Percent of time CGM glucose levels were between 70-180 mg/dl
% CGM >180 mg/dl | 72 hours
  Percent of time CGM glucose levels were >180 mg/dl
% CGM >250 mg/dl | 72 hours
  Percent of time CGM glucose levels were >250 mg/dl
number of SMBG <70 mg/dl | 72 hours
  Number of self monitored blood glucose levels less than 70 mg/dl
number of SMBG <60 mg/dl | 72 hours
  Number of self monitored blood glucose levels less than 60 mg/dl
number of SMBG <50 mg/dl | 72 hours
  Number of self monitored blood glucose levels less than 50 mg/dl
Grams of carbs for hypoglycemia | 72 hours
  Number of carbohydrates consumed for treatment of hypoglycemia
Total daily dose of insulin | 72 hours
  Total daily dose of insulin
% time CGM used | 72 hours
  Percent of time CGM was used
% time in closed loop | 72 hours
  Percent of time in closed loop
% of subjects with mean CGM <169 (eHbA1C < 7.5%) | 72 hours
  Percentage of subjects with mean CGM value < 169 for the 72 hour period. This corresponds to an estimated hemoglobin A1c of <7.5%.

OTHER OUTCOMES:
Comparison of Announced and Unannounced Meals | 72 hours
  Glycemic control in the 4 hour period after announced meals will be compared to glycemic control in the 4 hour period after unannounced meals as an exploratory measure
Safety Criteria 1: No more than 3 SMBG values < 50 mg/dL per subject | 72 hours
  Safety evaluation of system based on SMBG detected severe hypoglycemia
Safety Criteria 2: No more than 2 episodes with SMBG value >300 mg/dL for >1 hour not due to infusion set failure per subject | 72 hours
  Safety evaluation of system based on SMBG detected hyperglycemia
Safety Criteria 3: No kotonemia >1.0 mmol/L, while the system is functional unless related to an intercurrent illness or infusion set failure for any patient | 72 hours
  Safety evaluation of system based on ketone detection
Safety Criteria 4: No seizures or loss of consciousness while system is on and functional | 72 hours
  Safety evaluation of system based on severe hypoglycemic events

IPD SHARING:
Plan to Share IPD: No